CLINICAL TRIAL: NCT00081627
Title: COFU: A Multi-Center Phase II Clinical Trial to Evaluate the Safety and Efficacy of Weekly Treatment With CoFactor and 5-Fluorouracil in Patients With Metastatic Colorectal Carcinoma
Brief Title: Clinical Trial in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-CoFactor
Record Dates: First submitted 2004-04-15; First posted 2004-10-14 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — 5,11-methenyltetrahydrohomofolate; Fluorouracil

INTERVENTIONS:
Drug: CoFactor and 5FU

SUMMARY:
The objectives of this trial are to determine if CoFactor in combination with 5-FU are effective in the treatment of metastatic colorectal cancer and to determine the side effects observed with the administration of CoFactor and 5-FU.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have surgically incurable colon or rectal adenocarcinoma
* Karnofsky Performance Status of 60% or greater
* Patients may have symptomatic neuropathy
* Patients must have a life expectancy of at least 4 months
* Patients must be alimenting, receiving at least 1500Kcal/day nutrition, by any route
* Patients must have bidimensional measurable disease for response assessment
* Patients may have received adjuvant chemotherapy with fluoropyrimidine therapy
* Patients must have recovered from the toxicities of prior therapy, at least 4 weeks since prior adjuvant chemotherapy and major surgery
* Serum creatinine less than 2.4mg%, serum bilirubin less than 3.0mg%, WBC greater than 3,200/mm2, AGC greater than 1,500/mm3, platelet count greater than 90,000/mm3 and SGOT (AST) and SGPT (ALT) less than 3 times the upper limit of normal
* Male and non-pregnant, non-lactating female patients must be >18 years old.

Exclusion Criteria:

* Concurrent infection
* Failure of the patient or the patient's legal representative to sign the Informed consent
* Inability to obtain Informed Consent because of psychiatric or complex medical problem
* Patients with unstable oncologic emergency
* Patients with unstable medical conditions such as angina, transient ischemic attacks, rising creatinine, accelerated hypertension, etc.
* Cerebellar neurologic syndromes such as Parkinson's Disease, multiple sclerosis and amyotonia
* Known intolerance to fluoropyrimidine therapy suggestive of dihydropyrimidine dehydrogenase deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-04; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Reid, MD, PhD, Principal Investigator — University of California, San Diego
Locations (9):
- United States (5):
  - UCSD Moores Cancer Center, La Jolla, California
  - Mercy General Hospital, Sacramento, California
  - VA San Diego Healthcare System, San Diego, California
  - Spectrum Health, Grand Rapids, Michigan
  - Killeen Cancer Center, Killeen, Texas
- Serbia and Montenegro (4):
  - CHC Bezanijska Kosa, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Institute for Oncology and Radiology Serbia, Belgrade
  - Institute of Oncology, Sremska Kamenica